CLINICAL TRIAL: NCT06383403
Title: A Phase IIIb Randomised, Parallel-Group, Double-Blind, Placebo-Controlled, Two-Arm Study to Evaluate the Effect of Elafibranor 80 mg on Normalisation of Alkaline Phosphatase in Adult Participants With Primary Biliary Cholangitis (PBC) and Inadequate Response or Intolerance to Ursodeoxycholic Acid.
Brief Title: A Study of Elafibranor in Adults With Primary Biliary Cholangitis and Inadequate Response or Intolerance to Ursodeoxycholic Acid.
Acronym: ELSPIRE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-60190-463; 2024-510695-20-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elafibranor 80 mg (Experimental): Participants will take 1 tablet of elafibranor 80 mg per day orally before breakfast with a glass of water at approximately the same time each morning.
  Interventions: Drug: Elafibranor
- Placebo (Placebo Comparator): Participants will take 1 placebo tablet per day orally before breakfast with a glass of water at approximately the same time each morning.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Elafibranor — Round and orange film coated tablet of 80 mg.
  Other Names: IPN60190
  Arms: Elafibranor 80 mg
Other: Placebo — Round and orange film coated tablet of placebo
  Arms: Placebo

SUMMARY:
The participants in this study will have confirmed PBC with inadequate response or intolerance to Ursodeoxycholic acid (UDCA), which is a medication used in the management and treatment of cholestatic liver disease.

Primary biliary cholangitis is a slowly progressive disease characterised by damage of the bile ducts in the liver, leading to a build-up of bile acids which causes further damage. The liver damage in PBC may lead to scarring (cirrhosis). PBC may also be associated with multiple symptoms.

Many patients with PBC may require a liver transplant or may die if the disease progresses and a liver transplant is not done. This study will compare a daily dose of elafibranor (the study drug) to a daily dose of placebo (a dummy treatment).

The main aim of this study is to determine if elafibranor is better than placebo in reducing ALP levels to a normal value. High ALP levels in the blood can indicate liver disease.

There will be three periods in this study: A screening period (up to 8 weeks) to assess whether the participant can take part; a treatment period (up to 52 weeks) where eligible participants will be grouped as per their blood ALP levels and randomly assigned to either receive elafibranor or placebo, and a follow-up period (4 weeks) where participants' health will be monitored.

Participants will be twice as likely to receive elafibranor than placebo (2:1 ratio).

Participants will undergo blood sampling, urine collections, physical examinations, clinical evaluations, electrocardiograms (ECG: recording of the electrical activity of heart), ultrasound examinations (a noninvasive test that passes a probe over skin to look at the bladder, urinary tract, and liver), and Fibroscan® examinations (a noninvasive test that passes a probe on skin to measure stiffness of the liver).

They will also be asked to fill in questionnaires. Each participant will be in this study for up to 64 weeks (15 months).

ELIGIBILITY:
Inclusion Criteria

* Male or female participants age ≥18 years of age.
* Participants with a historical diagnosis of PBC as demonstrated by the presence of ≥2 of the following three historical diagnostic criteria:

  * i. History of elevated ALP levels for ≥6 months prior to the first screening visit (SV1).
  * ii. Positive Antimitochondrial antibody (AMA) titres (≥1/40 on immunofluorescence or M2 positive by enzyme linked immunosorbent assay) or positive PBC-specific antinuclear antibodies.
  * iii. Liver biopsy consistent with PBC.
* ALP >1 × ULN and <1.67 × ULN.
* Participants taking UDCA should have been on this medication for at least 6 months and at a stable dose for ≥3 months. Participants who are intolerant to UDCA should have taken the last dose of UDCA ≥3 months prior.
* Participants taking medications for management of pruritus must be on a stable dose for ≥3 months.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies

  * (a) Male participants must agree that, if their partner is at risk of becoming pregnant, they will use an effective method of contraception. The participant must agree to use contraception during the whole period of the study and for 30 days after the last dose of study intervention.
* Capable of giving signed informed consent

Exclusion Criteria

* History or presence of other concomitant liver diseases.
* Participants with known cirrhosis who have a Child-Pugh B or C score. Participants with cirrhosis with Child-Pugh A score are allowed.
* History of liver transplantation.
* History or presence of clinically significant hepatic decompensation.
* Known history of human immunodeficiency virus (HIV) infection.
* Medical conditions that may cause non-hepatic increases in ALP (e.g. Paget's disease).
* Evidence of any other unstable or untreated clinically significant conditions that are not well controlled.
* Medical condition with a life expectancy <2 years.
* Known malignancy or history of malignancy within the last 2 years, except for successfully treated localised basal cell carcinoma or squamous cell carcinoma of the skin; or in-situ carcinoma of the uterine cervix.
* History of hepatocellular carcinoma.
* Alpha-foetoprotein (AFP) >20 ng/mL with 4-phase liver computed tomography (CT) or magnetic resonance imaging (MRI) scans suggesting presence of liver cancer.
* Administration of the following medications is prohibited during the study, and prior to the study as per the timelines specified below:

  * i. Systemic (oral or parenteral) use within 3 months prior to SV1 of: fibrates, seladelpar, glitazones, obeticholic acid, azathioprine, cyclosporine, methotrexate, mycophenolate, or long-term systemic corticosteroids (parenteral and oral chronic administration only); potentially hepatotoxic drugs (including α-methyl-dopa, valproic acid, isoniazid or nitrofurantoin)
* Participants with previous exposure to elafibranor.
* Participants who are currently participating in, plan to participate in, or have participated in an investigational drug study or medical device study containing active substance within 30 days or 5 half-lives, whichever is longer.
* Total bilirubin (TB) >2 × ULN. Participants with Gilbert's syndrome are eligible with a TB above 2 × ULN if direct bilirubin is <30% of TB.
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >5 × ULN.
* Creatine phosphokinase (CPK) >2 × ULN.
* Platelet count <75,000/µL.
* International normalised ratio >1.3 in the absence of anticoagulant therapy.
* Estimated glomerular filtration rate (eGFR) <45 mL/min/1.73m2.
* Significant renal disease, including nephritic syndrome, chronic kidney disease (defined as participants with evidence of significantly impaired kidney function or underlying kidney injury).

Other exclusions

* For female participants: known pregnancy, or has a positive serum pregnancy test, or is breastfeeding.
* Regular alcohol intake in excess of the recommended limit of 2 standard drinks per day for men or 1 standard drink per day for women.
* History of alcohol abuse, or other substance abuse within 1 year prior.
* Known hypersensitivity to the investigational product or to any of the excipients of elafibranor.
* Mental instability or incompetence, such that the validity of informed consent or ability to be compliant with the study is uncertain.
* Any other condition that, in the opinion of the investigator, would interfere with study participation or completion, or would put the participant at risk, including a potential participant assessed as being at high risk of noncompliance with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-06-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with normalisation of Alkaline Phosphate (ALP) Levels | At Week 52

SECONDARY OUTCOMES:
Percentage of participants with normalisation of ALP Levels | From baseline to Week 4, Week 12, Week 24 and Week 36
Change from baseline in ALP levels | From baseline to Week 4, Week 12, Week 24, Week 36 and Week 52
Percentage of participants with normalisation of ALP Levels and ≥15% decrease from Baseline | From baseline to Week 4, Week 12, Week 24, Week 36 and Week 52
Percentage of participants with ≥40% decrease from Baseline in ALP Levels | From baseline to Week 4, Week 12, Week 24, Week 36 and Week 52
Percentage of participants with ALP <0.5 × Upper Limit of Normal (ULN) | At Week 4, Week 12, Week 24, Week 36 and Week 52
Changes from baseline in Total Bilirubin (TB) Levels | From baseline to Week 4, Week 12, Week 24, Week 36 and Week 52
Percentage of participants with TB <0.7 × ULN | At Week 4, Week 12, Week 24, Week 36 and Week 52
Percentage of participants with normalisation of ALP and TB <0.7 × ULN | At Week 4, Week 12, Week 24, Week 36 and Week 52
Percentage of participants with normalisation of TB and ALP Levels | At Week 4, Week 12, Week 24, Week 36 and Week 52
Percentage of participants with complete biochemical response | At Week 4, Week 12, Week 24, Week 36 and Week 52
  Defined as normal levels of TB, ALP, aminotransferases, albumin, and International normalised ratio (INR)
Change from baseline in PBC Worst Itch Numeric Rating Scale (NRS) score | From baseline through Week 52
  PBC Worst Itch Numeric Rating Scale (NRS) is a self-administered patient-reported outcome questionnaire that measures itch intensity. It asks participants to rate the intensity of their Worst Itch on an 11-point scale ranging from 0 (no itch) to 10 (Worst Itch imaginable): - once daily (24-hour recall period)
Percentage of participants with moderate to severe pruritus at baseline (i.e. score ≥4) with a clinically meaningful response in PBC Worst Itch NRS | From baseline through Week 52
  Defined as ≥1.8-point reduction from baseline
Change from baseline in 5-D itch score | From baseline to Week 4, Week 24, and Week 52
  Change from baseline in symptoms in terms of 5 domains: degree, duration, direction, disability and distribution. Patients rate their symptoms over the preceding 2-week period on a 1 to 5 scale, with 5 being the most affected.
Change from baseline in Patient Global Impression of Severity (PGI-S) scores | From baseline to Week 4, Week 24, and Week 52
  Patient Global Impression of Severity (PGI-S) is a 1-item, 5-point scale designed to assess the participant's impression of itch severity over the past 7 days, at different time points during the study.
Patient Global Impression of Change (PGI-C) scores | At Week 4, Week 24, and Week 52
  Patient Global Impression of Change (PGI-C) is a 1-item, 5-point scale designed to assess the participant's impression of change in itch severity since the baseline visit
Change from baseline in PBC-40 Quality of Life (QoL) scores | From baseline to Week 4, Week 24, and Week 52
  PBC-40 Quality of Life (QoL) assesses symptoms across six domains: fatigue, emotional, social, cognitive function, general symptoms and itch. Patients respond on a verbal response scale, depending on the section options range from 'never' / 'not at all' / 'strongly disagree' to 'always' / 'very much'/ 'strongly agree'. Five items (3/3 in the itch domain and 2/10 in the social domain) also include a 'does not apply' option. A score for each domain is provided (but a total score is not calculated), with each verbal response scale correlating to a score of 1-5 per item (0-5 on items with a 'does not apply' option) with 5 being the most affected. The PBC-40 has a 4-week recall period.
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form 7a scores | From baseline to Week 4, Week 24, and Week 52
  PROMIS Fatigue Short Form 7a scores consists of 7 items that measure both the experience of fatigue and the interference of fatigue on daily activities over the past week. Response options are on a 5-point Likert scale, ranging from 1 to 5. Scores can range from 7 to 35, with higher scores indicating greater fatigue.
Percentage of participants experiencing Treatment- Emergent Adverse Events (TEAEs), treatment- related TEAEs, Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs). | From baseline until 4 weeks after the end of treatment (maximum duration of 52 weeks)
  An Adverse Event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AESIs are AEs that may not be serious but are of special importance to a particular drug or class of drugs.
Percentage of participants developing clinically significant changes in physical examination | From baseline until 4 weeks after the end of treatment (maximum duration of 52 weeks)
  The clinical significance will be graded by the investigator.
Percentage of participants developing clinically significant changes in vital signs | From baseline until 4 weeks after the end of treatment (maximum duration of 52 weeks)
  The clinical significance will be graded by the investigator.
Percentage of participants developing clinically significant changes in Electrocardiogram (ECG) Readings | From baseline until 4 weeks after the end of treatment (maximum duration of 52 weeks)
  The clinical significance will be graded by the investigator.
Percentage of participants developing clinically significant changes in laboratory parameters | From baseline until 4 weeks after the end of treatment (maximum duration of 52 weeks)
  The following laboratory parameters will be reported: blood chemistry, hematology and coagulation, liver tests and renal tests (including urinalysis). The clinical significance will be graded by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (60):
- United States (20):
  - Southern California Research Center, Coronado, California
  - Topgraphy Health, Inc., Los Angeles, California
  - University of California, Davis, Sacramento, California
  - Stanford University Medical Center, Stanford, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Rocky Mountain Gastroenterology, Littleton, Colorado
  - International Center for Research, Tampa, Florida
  - Delta Research Partners, LLC, West Monroe, Louisiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - Huron Gastroenterology Associates - Center for Digestive Care, Ypsilanti, Michigan
  - South Denver Gastroenterology,P.C., Englewood, New Jersey
  - Southwest Gastroenterology Associates, PC (SWGA), Albuquerque, New Mexico
  - Northwell Health Center for Liver Disease and Transplantation, Manhasset, New York
  - Charlotte Gastroenterology & Hepatology, PLLC, Charlotte, North Carolina
  - Coastal Research Institute, Fayetteville, North Carolina
  - Gastroenterology Center of the Midsouth, Cordova, Tennessee
  - Methodist Transplant Physicians, Dallas, Texas
  - American Research Corporation at The Texas Liver Institute, San Antonio, Texas
  - American Research Corporation, San Antonio, Texas
  - Velocity Liver Institute NW, Seattle, Washington
- Czechia (4):
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Artroscan, Ostrava
  - Research Site s.r.o., Pilsen
  - Institute for Clinical and Experimental Medicine - IKEM, Prague
- Clinique Pasteur, Toulouse, France
- Germany (4):
  - Universitatsklinikum Heidelberg, Heidelberg
  - Gastroenterologsiche Studiengesellschaft Herne, Hemer
  - EUGASTRO GmbH, Leipzig
  - Universitaetsklinikum Muenster, Münster
- Italy (4):
  - Ospedale Policlinico San Martino - IRCCS, Genova
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - IRCCS Istituto clinico humanitas - Humanitas Mirasole spa, Rozzano
- Poland (2):
  - Krakowskie Centrum Medyczne Sp.z.o.o - FutureMeds, Krakow
  - FutureMeds Warszawa Centrum, Warsaw
- Romania (2):
  - Cluj County Clinical Emergency Hospital, Cluj-Napoca
  - Gastromedica Srl, Iași
- South Korea (10):
  - Korea University Ansan Hospital, Ansan-si
  - Keimyung University Dongsan Hospital, Daegu
  - Kyungpook National University Hospital (KNUH), Daegu
  - Pusan National University Hospital (PNUH), Pusan
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Seoul National University Bundang Hospital (SNUBH), Seongnam-si
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
- Spain (6):
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda
  - Institut d Investigacio i Innovacio Parc Tauli, Hospital Universitari Parc Tauli, Sabadell
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (7):
  - Aberdeen Royal Infirmary NHS Grampian Grampian Health Board, Aberdeen
  - Bradford Royal Infirmary - Bradford Teaching Hospitals NHS Foundation, Bradford
  - Frimley Park Hospital - Frimley Health NHS Foundation Trust, Frimley
  - Queen Elizabeth University Hospital - Greater Glasgow Health Board, Glasgow
  - Hull Royal Infirmary - Hull University Teaching Hospitals NHS Trust, Hull
  - Ambrose King Centre-Royal London Hospital-Barts Health NHS Trust, London
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/